CLINICAL TRIAL: NCT01456520
Title: An Open Label, Single Dose, Randomized, Two-Period, Two-Way Crossover Study to Evaluate the Pharmacokinetics and Bioequivalence of Vycavert Tablets Compared to Norco® Tablets in Healthy Subjects
Brief Title: Pharmacokinetics and Bioequivalence of Vycavert (10 mg Hydrocodone Bitartrate/325 mg Acetaminophen) Compared to the Reference Drug Norco
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4571001
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: pharmacokinetics; bioequivalence; hydrocodone; acetaminophen; moderate to moderately severe pain
MeSH Terms: interventions — oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: single dose Vycavert (Test) (Experimental)
  Interventions: Drug: Vycavert
- B: single dose Norco (Reference) (Active Comparator)
  Interventions: Drug: Norco

INTERVENTIONS:
Drug: Vycavert — single dose Vycavert containing 10 mg hydrocodone bitartrate/325 mg acetaminophen
  Arms: A: single dose Vycavert (Test)
Drug: Norco — single dose Norco containing 10 mg hydrocodone bitartrate/325 mg acetaminophen
  Arms: B: single dose Norco (Reference)

SUMMARY:
This study aims to determine whether the hydrocodone and acetaminophen exposures following oral dosing of Vycavert are comparable to those following oral dosing of Norco.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant disease
* History of obstructive sleep apnea
* Life time history and/or recent evidence of alcohol and/or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) to time infinity (inf) (if data permit), otherwise (AUC) to last quantifiable concentration (last) of hydrocodone. | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
Area Under the Curve (AUC) to time infinity (inf) (if data permit), otherwise (AUC) to last quantifiable concentration (last) of acetaminophen | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
Cmax (maximum plasma concentration) of of hydrocodone | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
Cmax (maximum plasma concentration) of acetaminophen | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose

SECONDARY OUTCOMES:
AUClast of hydromorphone and norhydrocodone | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
Cmax of hydromorphone and norhydrocodone | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
T1/2 (half life) as data permit of hydrocodone, hydromorphone, norhydrocodone, and acetaminophen | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
Tmax (Time at maximum concentration) of hydrocodone, hydromorphone, norhydrocodone, and acetaminophen | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose
Adverse events, vital signs, pulse oximetry and laboratory parameters. | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4571001&StudyName=Pharmacokinetics%20and%20Bioequivalence%20of%20Vycavert%20%2810%20mg%20Hydrocodone%20Bitartrate/325%20mg%20Acetaminophen%29%20Compared%20to%20the%20Reference%20Drug%20Norco